CLINICAL TRIAL: NCT06173700
Title: Empowering Parental Caregivers: A Virtual Support Group With Problem Solving Training for Parents/Guardians of Children With SCI/D
Brief Title: Empowering Parental Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duquesne University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2023/04/8
Record Dates: First submitted 2023-11-30; First posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-11

CONDITIONS: Caregivers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Group Intervention (Experimental): 7-week web-based group with problem solving training
  Interventions: Behavioral: web-based group problem solving and coping training

INTERVENTIONS:
Behavioral: web-based group problem solving and coping training — The group included one-hour, weekly Zoom sessions, that were facilitated by an occupational therapy doctoral candidate (first author) for 7 consecutive weeks. During the first session, the candidate explained adaptive and maladaptive coping strategies and asked each participant to identify one adaptive coping strategy that they currently use and will continue to use in the future. The candidate then explained the FOCUS problem-solving approach. For each session afterward, the candidate presented a topic-related scenario for parents to identify an effective solution using the FOCUS steps (APA, 2011). Parent-chosen topics included recreation, assistive technology, motivating and advocating, physical activity, skin integrity, and adaptive fashion. The general process of the meetings is presented in Figure 1. After every meeting the candidate sent out a summary of resources that were discussed during the meeting, ultimately putting them all together in an "Empowering Caregiver Guide."

SUMMARY:
The goal of this clinical trial was to learn about the feasibility and pilot outcome measures in caregivers of children with spinal cord injury who completed a 7-week problem-solving training web-based group. The main question it aims to answer is: What is the feasibility of a seven-week, occupational therapist-facilitated, web-based support group with problem-solving training for parental caregivers of children with SCI?

Participants participated 1 time a week for seven weeks in a web-based group group:

* learning about the FOCUS problem-solving model
* applying positive coping and problem-solving strategies to current issues.

ELIGIBILITY:
Inclusion Criteria:

* one must be a parent or guardian of a child with a spinal cord injury or disorder, be that child's primary caregiver, and be 18 years or older.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-06-06 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-08-09 (Actual)

PRIMARY OUTCOMES:
Brief COPE | Before the group began, 7 weeks after start of group
  The Brief COPE is a 28-item self-report measure that determines the participants' styles of coping (Carver,1997).
Caregiver Self-Assessment Questionnaire | Before the group began 7 weeks after start of group
  The Caregiver Self-Assessment Questionnaire is a brief, 18-question self-assessment that asks respondents to consider the impact of caregiving on their stress levels, physical body, and mental health (American Society for Geriatrics, 2015).
Knowledge Check | Before the group began 7 weeks after start of group
  The Knowledge Check was a measure developed by the research team with guidance from Obst and Porter's guide for school personnel (n.d.). The research team generated the items around three themes: general SCI knowledge, FOCUS problem-solving skills, and coping knowledge.

SECONDARY OUTCOMES:
Attendance | across the 7 weeks of the group
  number of sessions attended
Client Satisfaction Questionnaire-8 (CSQ-8) | at the end of the 7 weeks
  The CSQ-8 is an eight-item standardized questionnaire that aims to understand the participants' general satisfaction with the sessions, developed by Attkisson & Greenfield (2004). It is a highly effective tool to measure client satisfaction with program contents and has high internal consistency (Attkisson & Greenfield, 2004).

CONTACTS AND LOCATIONS:
Overall Officials: Elena Donoso Brown, PhD, Study Chair — Duquesne University; Elena Martino, BS, Principal Investigator — Duquesne University
Locations (1):
- United Spinal Association, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No